CLINICAL TRIAL: NCT00001806
Title: Methods in Education for Breast Cancer Genetics
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 990081; 99-C-0081; NCT00019877 (obsolete NCT alias)
Record Dates: First submitted 1999-11-03; First posted 1999-11-04 (Estimated); Last update posted 2019-12-12 (Actual); Status verified 2017-12-06

CONDITIONS: Breast Cancer; Ovarian Cancer
Keywords: Genetic Testing; Genetic Counseling; BRCA1/BRCA2; Genetic Education; Informed Consent; Breast Cancer; Ovarian Cancer; Known Family Mutation
MeSH Terms: conditions — Breast Neoplasms; Ovarian Neoplasms; Fanconi Anemia, Complementation Group D1 | interventions — Counseling

ARMS (2):
- Group (Experimental): Group education and counseling
  Interventions: Other: Genetic Education and Counseling
- Individual (Active Comparator): Individual education and counseling
  Interventions: Other: Genetic Education and Counseling

INTERVENTIONS:
Other: Genetic Education and Counseling — Group Education and Counseling
  Arms: Group
Other: Genetic Education and Counseling — Individual Education and Counlseing
  Arms: Individual

SUMMARY:
In 1997, the Genetics Department of the NCI Medicine Branch helped establish a breast cancer genetics program at the National Naval Medical Center s Breast Care Center. Genetic education, counseling, and germline testing for BRCA1 and BRCA2, two genes which confer increased lifetime risks for breast and ovarian cancer, were offered under a Navy IRB-approved study. Sixty participants received education and counseling on that protocol, 49 of whom chose to have genetic testing. The education and counseling, provided by oncology nurses trained in cancer genetics, focused on preparing participants to make well-informed decisions about testing. Included were information on cancer and genetics; hereditary breast/ovarian cancer syndrome; risks, benefits and limitations of BRCA1/BRCA2 testing; and screening and risk reduction options for high-risk individuals. Through our experience with this study, we devised two different methods of providing this information. Both of these methods were well received and appear to be equally effective, as measured by knowledge assessments before and after the sessions and subjective evaluation by the participants. We will now study them in a randomized fashion in the current protocol, to better evaluate whether one method is preferable. Ultimately we hope to be able to make recommendations that will allow for access to genetic education and counseling for more individuals in a more cost efficient manner.

DETAILED DESCRIPTION:
In October 1995 the National Naval Medical Center opened the only Department of Defense funded Breast Care Center (BCC). Within less than one year the Center was seeing 100 - 200 new patients per week and making 10 - 20 new diagnoses of breast cancer per month. In 1997 we began conducting germline testing for BRCA1 and BRCA2 under an approved Navy IRB study. To date, 51 individuals have enrolled into the Education and Counseling component, and 42 individuals have elected to receive germline testing. Early on it became apparent that a more time efficient approach to education and counseling would be required if access to information on breast cancer genetics was to be made available to a larger population. Traditionally, education and counseling has been offered on a one to one basis prior to germline testing. Often, hours are spent with an individual. At some centers, multiple visits are standard. Not only is there a shortage of health care providers trained in cancer genetics, but even if there were an abundance of trained providers, the time and cost, as well as need for efficiency would preclude this type of approach. Thus, this approach is not applicable to most health care delivery systems. We began offering education in small groups approximately 18 months ago, using the same informational content that we use in our one to one sessions. Based on preliminary, nonrandomized results, there appeared to be no difference in learning and general patient satisfaction based on results of pre- and post-test administered before and after the education. It was our contention that group education is equivalent, and in some situations better than individual education. Therefore, we will conduct a randomized trial designed to test equivalence between individual and group education.

ELIGIBILITY:
* INCLUSION CRITERIA:

At least one of the following:

Diagnosis of breast cancer, or DCIS prior to or at 45, or ovarian cancer prior to or at age 50;

Diagnosis of breast cancer with bilateral disease or multiple primaries or breast cancer and ovarian cancer in the same individual;

Diagnosis of breast or ovarian cancer and one first or second degree relative with breast cancer diagnosed prior to or at age 45, or ovarian cancer prior to or at age 50;

Diagnosis of breast or ovarian cancer and three relatives in the same lineage with breast or ovarian cancer; each affected individual must be a first- or second-degree relative to another of the affected individuals;

Diagnosis of breast or ovarian cancer and a first or second degree male relative with breast cancer;

A woman of Ashkenazi Jewish descent who meets any of the above criteria, with specified ages of onset of 50 for breast cancer and any age for ovarian cancer;

A male with breast cancer diagnosed at any age;

Documented BRCA mutation in the family.

All individuals must be able to give informed consent.

EXCLUSION CRITERIA:

Patients will be considered ineligible for any of the following reasons:

Any psychological disorder which may hinder the participant's ability to understand and process the material, based on a psychiatric consultation.

Inable to return for 2 visits.

Age under 18 years old.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Actual)
Dates: Start 1999-04-06; Primary Completion 2017-12-06 (Actual); Study Completion 2017-12-06 (Actual)

PRIMARY OUTCOMES:
Impact of Events Scale | Baseline, 3, 6, and 12 months
Breast Cancer Genetics Knowledge Score | Baseline, 3, 6, and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen Calzone, R.N., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- Walter Reed National Medical Center, Bethesda, Maryland, United States

REFERENCES:
- [Background] Statement of the American Society of Clinical Oncology: genetic testing for cancer susceptibility, Adopted on February 20, 1996. J Clin Oncol. 1996 May;14(5):1730-6; discussion 1737-40. doi: 10.1200/JCO.1996.14.5.1730. PMID 8622094
- [Background] Statement of the American Society of Human Genetics on genetic testing for breast and ovarian cancer predisposition. Am J Hum Genet. 1994 Nov;55(5):i-iv. No abstract available. PMID 7977337
- [Background] Hoskins KF, Stopfer JE, Calzone KA, Merajver SD, Rebbeck TR, Garber JE, Weber BL. Assessment and counseling for women with a family history of breast cancer. A guide for clinicians. JAMA. 1995 Feb 15;273(7):577-85. PMID 7837392